CLINICAL TRIAL: NCT00678860
Title: Pilot Validation Study of Computer Administration of Vision Targeted Quality of Life Instruments
Brief Title: Validation of Computerized Vision-Targeted Quality-of-Life Questionnaires
Status: Completed | Type: Observational
Sponsor: National Eye Institute (NEI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 080135; 08-EI-0135
Record Dates: First submitted 2008-05-14; First posted 2008-05-16 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-10-31

CONDITIONS: Eye Disease
Keywords: Questionnaire; Computer Assisted Interface; Quality of Life; Dry Eye; Ocular Surface Disease; Healthy Volunteer; HV
MeSH Terms: conditions — Eye Diseases; Dry Eye Syndromes

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This study will test and compare computerized and paper versions of eye questionnaires. Questionnaires are used in medicine to gain a better understanding of how a disease can impact a person's quality of life. Computerized versions of such questionnaires are often as good as or better than paper versions, but there has been no direct comparison of the two. This study may help in the development of eye questionnaires used to understand symptoms and monitor patients in clinical trials.

People 21 years of age and older with ocular surface disease (OSD) and matched control subjects without OSD may be eligible for this study. All participants undergo the following procedures:

* Medical and eye history.
* Vision test and examination of the front part of the eye.
* Tear measurement: A small piece of paper is placed on the surface of the eye to measure the amount of tears produced. The consistency of the tears is measured by looking at how fast they evaporate from the surface of the eye.
* Completion of either paper-based or computer-based version of a questionnaire 15 minutes after the eye examination and completion of the other version within 1 week at home. (Subjects who complete the paper version in the clinic are told how to access the computer version online at home or on a library computer; those who complete the computer version in the clinic are given a paper version to take home.)

DETAILED DESCRIPTION:
The purpose of this protocol is to compare the health-related quality of life (visual function) reported by participants when using web-based questionnaires versus their responses obtained when using standard paper versions of the questionnaires. This comparison will be performed in a population of patients diagnosed with ocular surface disease (OSD) and in age- and gender-matched controls by using a randomized, cross-over study design. This type of comparative study of patient-reported outcomes has been reported for rheumatology, cardiology, psychiatry, asthma, alcoholism, pain assessment, gastrointestinal disease, diabetes, and allergy populations; however, to our knowledge there have been no reports of such a study from patients with ocular disease. The study will evaluate the agreement between scores reported via two modes of administration: a web-based version and a paper-and-pencil version. Components of three questionnaires commonly used to evaluate visual function, symptoms, and vision-related quality of life in OSD will be included: the initial 5 questions of the Ocular Surface Index (OSDI), question #15 of the National Eye Institute Visual Functioning Questionnaire - 25 (VFQ-25), and specified domains of the National Eye Institute Refractive Error Quality Of Life Instrument-42 (RQL-42) (clarity of vision, near vision, far vision, glare, symptoms, worry, and satisfaction with correction).

The study will also evaluate whether there are differences in mean overall score by age, gender, order of administration, or disease severity.

Ocular surface disease, which includes dry eye disease secondary to a variety of etiologies, is an ophthalmic condition which places a burden not just on functional vision, but also on overall health related quality of life (HRQoL), with an impact similar to that of moderate angina3. This study will add to the body of knowledge in the field of patient-reported outcome measures (PROs), and will be the first to compare the computerized, web-based and paper-based versions of previously validated questionnaires used to assess QoL in subjects with ocular disease.

There has been an increasing interest in assessing PROs in many fields of medicine, especially in the context of clinical trials where HRQoL is an important component of the overall evaluation of an intervention or treatment. As the use of computers increases and accessibility to the internet broadens, there is a tremendous potential in harnessing this technology in the future as a cost-effective, efficient way to gather clinical data on PROs for future ophthalmic clinical trials and studies.

ELIGIBILITY:
* INCLUSION CRITERIA:

The study cohort will be comprised of eighty (80) participants diagnosed with OSD and 40 controls without OSD comprised of similar numbers of men and women.

INCLUSION CRITERIA FOR OSD GROUP:

* Patients greater than or equal to 18 years of age with a diagnosis of ocular surface disease confirmed by investigator.
* Schirmer I less than 10 mm wetting over 5 minutes OR tear breakup time less than or equal to 5 seconds.
* Binocular visual acuity at near equal to or greater than 20/40 (Jaeger 3) with habitual correction.
* Literacy and fluency in English sufficient to follow study instructions and likely to be able to comprehend the questionnaires.
* Ability and willingness to complete the study protocol.

EXCLUSION CRITERIA FOR OSD GROUP:

* Ocular surgery or infection within 3 months of study enrollment.
* Inability to obtain appropriate consent.
* Allergy or sensitivity to any medication used in study.
* Subject has a situation or condition, which in the investigator's opinion, may put the subject at a significant risk, may confound the study result, or may interfere significantly with the participation in the study.
* Uncontrolled systemic disease.
* Active ocular disease other than ocular surface disease which in the investigator's opinion may put the subject at a significant risk, may confound the study result, or may interfere significantly with the participation in the study.
* Any disability preventing timely, efficient completion of writing or keyboarding tasks.
* Incapable of providing informed consent.
* Monocular vision (legal blindness in one eye).

INCLUSION CRITERIA FOR CONTROL GROUP:

* Age greater than or equal to 18 years.
* Schirmer I test greater than or equal to 10 mm wetting over 5 minutes OR tear breakup time greater than 5 seconds.
* Binocular visual acuity at near equal to or greater than 20/40 (Jaeger 3) with habitual correction
* Literacy and fluency in English sufficient to follow study instructions and likely to be able to comprehend the questionnaire
* Ability and willingness to complete the study protocol

EXCLUSION CRITERIA FOR CONTROL GROUP:

* A diagnosis of ocular surface disease made by a clinician
* Ocular surgery or infection within 6 months of study enrollment
* Pupillary, motility, convergence or accommodative ocular disorder judged by investigator to have potential to negatively impact ease of near and intermediate binocular visual function
* Inability to obtain appropriate consent
* Allergy or sensitivity to any medication used in study.
* Monocular vision (legal blindness in one eye) or subject has a situation or condition, which in the investigator's opinion, may put the subject at a significant risk, may confound the study results, or may interfere significantly with the participation in the study.
* Uncontrolled systemic disease
* Active ocular disease which in the investigator's opinion may put the subject at a significant risk, may confound the study result, or may interfere significantly with the participation in the study
* Any disability preventing timely, efficient completion of writing or keyboarding tasks

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2008-05-09; Study Completion 2011-10-31

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Study protocol for the World Health Organization project to develop a Quality of Life assessment instrument (WHOQOL). Qual Life Res. 1993 Apr;2(2):153-9. PMID 8518769
- [Background] Miljanovic B, Dana R, Sullivan DA, Schaumberg DA. Impact of dry eye syndrome on vision-related quality of life. Am J Ophthalmol. 2007 Mar;143(3):409-15. doi: 10.1016/j.ajo.2006.11.060. Epub 2007 Jan 2. PMID 17317388
- [Background] Schiffman RM, Walt JG, Jacobsen G, Doyle JJ, Lebovics G, Sumner W. Utility assessment among patients with dry eye disease. Ophthalmology. 2003 Jul;110(7):1412-9. doi: 10.1016/S0161-6420(03)00462-7. PMID 12867401